CLINICAL TRIAL: NCT06687668
Title: Short Leg Walking Plaster Cast Versus Walking Foot Cast for Jones Fracture: An Open Label Randomized Controlled Trial.
Brief Title: Short Leg Walking Plaster Cast Versus Walking Foot Cast for Jones Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/010
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Jones Syndrome; Metatarsal Bone Fractures
Keywords: Jones Fracture; Non-Surgical Management; Conservative Treatment; Walking Cast; Plaster Cast Treatment
MeSH Terms: conditions — Jones syndrome

STUDY DESIGN:
Intervention Model Description: Two arms in parallel: One group receives the Short Leg Walking Plaster Cast, and the other receives the Walking Foot Plaster Cast.
Masking Description: No masking due to the visible nature of the interventions (type of plaster cast), but the outcomes assessor is blinded to treatment assignment when evaluating follow-up outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Leg Walking Plaster Cast (Experimental): Participants in this group will receive a short leg walking plaster cast, extending from the metatarsal heads up to the mid-calf. This cast limits mobility at the fracture site while allowing partial weight-bearing as tolerated. Participants will use this cast for six weeks, with follow-up for fracture healing and functional outcome at the end of the treatment period.
  Interventions: Other: Short Leg Walking Plaster Cast
- Walking Foot Plaster Cast (Active Comparator): Participants in this group will receive a walking foot plaster cast, which provides support to the foot while allowing more flexibility around the ankle. This cast restricts movement to avoid further injury while enabling weight-bearing activities as tolerated. The cast will be worn for six weeks, with follow-up assessments for fracture healing and functional outcome after this period.
  Interventions: Other: Walking Foot Plaster Cast

INTERVENTIONS:
Other: Short Leg Walking Plaster Cast — A short leg walking plaster cast that extends from the head of the metatarsal to the mid-calf. This cast provides stability to the fracture site while allowing limited weight-bearing, and is designed to restrict inversion and eversion movements, thereby reducing the risk of fracture displacement. Applied for six weeks.
  Arms: Short Leg Walking Plaster Cast
Other: Walking Foot Plaster Cast — A walking foot plaster cast that covers the foot from the metatarsal heads but leaves the toes exposed. This cast allows weight-bearing while restricting side-to-side movement, providing support to the fracture area without immobilizing the ankle. It will be used for six weeks.
  Arms: Walking Foot Plaster Cast

SUMMARY:
This study is an open-label, randomized controlled trial comparing the effectiveness of two plaster cast methods-Short Leg Walking Plaster Cast and Walking Foot Plaster Cast-for treating Jones fractures, a common fracture at the base of the fifth metatarsal in the foot. This trial will be conducted at Lady Reading Hospital Peshawar. The study will evaluate differences in fracture healing and functional outcomes between these two treatment approaches. Findings from this trial may guide more evidence-based treatment protocols for Jones fractures, potentially improving patient mobility and recovery without requiring surgical intervention.

DETAILED DESCRIPTION:
Jones fractures represent 26.3% of fractures at the base of the fifth metatarsal and are commonly treated conservatively through various weight-bearing casts. The lack of consensus on the optimal casting method for Jones fractures necessitates further study, particularly given the absence of published guidelines. This trial, unique in its randomized and prospective approach within Pakistan, aims to compare Short Leg Walking Plaster Casts and Walking Foot Plaster Casts specifically for Jones fractures.

Patients meeting the inclusion criteria will be randomly assigned to one of the two treatment groups, with the primary endpoints being fracture healing (union) and functional outcomes at six weeks, assessed via radiographs and the American Orthopaedic Foot and Ankle Score (AOFAS). This study seeks to produce robust evidence to inform treatment guidelines, allowing patients, especially in low- and middle-income settings, to continue daily activities with minimal disruption during recovery.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* 18 years and above
* Jones fractures that are un-displaced or minimally displaced (less than 2 mm)
* Fractures presented within 7 days of injury

Exclusion Criteria:

* Significant foot swelling
* Open fractures
* Ipsilateral foot, ankle, or lower limb soft tissue pathology or fractures
* Pathological fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Fracture Union Rate | 6 weeks after cast application.
  Measurement of fracture healing defined by callus formation and obliteration of the fracture line in 2 out of 3 cortices (lateral, medial, plantar) on X-ray, and absence of pain and tenderness at the fracture site, assessed by a senior orthopedic consultant.
Delayed Union Rate | 6 weeks, with further assessment at 8 weeks if needed.
  Defined by insufficient callus in fewer than 2 cortices and persistent pain and tenderness at the fracture site. This assessment determines cases where additional casting or intervention may be necessary.
Nonunion Rate | 8 weeks post-cast application.
  Nonunion is confirmed if there is insufficient callus formation in fewer than 2 cortices, with persistent pain and tenderness at the fracture site.
Functional Outcome (American Orthopaedic Foot and Ankle Score - AOFAS) | 6 weeks after cast removal.
  Functional outcome assessed via the AOFAS scoring system, which includes pain (40 points), function (50 points), and alignment (10 points), with higher scores indicating better function.

SECONDARY OUTCOMES:
Complication | Throughout the study duration up to 8 weeks.
  Incidence of any complications, such as cast-related issues, skin irritation, or infection, during and after cast application.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Faaiz Ali Shah, Principal Investigator — Lady Reading Hospital, Pakistan
Locations (1):
- Lady Reading Hospital, Pakistan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan includes making anonymized individual participant data (such as baseline demographics, primary and secondary outcomes, and adverse event data) available to qualified researchers for the purpose of further analysis or replication of the study findings. This data will be shared upon reasonable request and for research purposes only.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication of the primary study results, anticipated within 6-12 months following study completion, and will be accessible for a period of 5 years.
Access Criteria: Researchers must submit a formal request to the study team, including a brief research proposal, purpose, and intended analysis of the data. Data access will be granted upon review and approval of the request to ensure ethical use of the data.

REFERENCES:
- [Background] Buskova K, Bartonicek J, Rammelt S. Fractures of the Base of the Fifth Metatarsal Bone: A Critical Analysis Review. JBJS Rev. 2021 Oct 21;9(10). doi: 10.2106/JBJS.RVW.21.00010. PMID 34673663
- [Background] de Ruijter MA, Yuan JZ, Derksen RJ. The Clinical Outcomes of Operative Treatment Versus Conservative Treatment for Dancer's Fractures: Protocol for a Retrospective Cohort Study. JMIR Res Protoc. 2022 Apr 5;11(4):e37171. doi: 10.2196/37171. PMID 35380544
- [Background] Park JY, Kim HN, Hyun YS, Park JS, Kwon HJ, Kang SH, Kim GL. Effect of Weight-Bearing in Conservative and Operative Management of Fractures of the Base of the Fifth Metatarsal Bone. Biomed Res Int. 2017;2017:1397252. doi: 10.1155/2017/1397252. Epub 2017 Dec 26. PMID 29441351